CLINICAL TRIAL: NCT05098717
Title: End-expiratory Trans-pulmonary Pressure Guided PEEP Titration in Patients With Pulmonary Fibrosis and UIP Pattern Undergoing Mechanical Ventilation
Acronym: ETROPON
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio11
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Mechanical Ventilation Pressure High
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UIP patients: Patients with pulmonary fibrosis and UIP pattern undergoing mechanical ventilation for acute respiratory failure
- ARDS patients: Patients with ARDS undergoing mechanical ventilation for acute respiratory failure

SUMMARY:
Patients with pulmonary fibrosis and associated usual interstitial pneumonia that require mechanical ventilation for acute respiratory failure experience poor clinical outcomes. This may be influenced by the unfavorable interaction between the fibrotic lung and the stress and strain stimuli generated during controlled ventilation. Although there is no consensus on how to ventilate these patients, much of the recommendations followed in clinical practice are taken from the experience on patients with acute respiratory distress syndrome. Among these, measuring the esophageal pressures and adjusting positive-end expiatory pressure to make trans-pulmonary pressures positive can decrease atelectasis, derecruitment of lung, and cyclical opening and closing of airways and alveoli, thus optimizing lung mechanics and oxygenation. The effect of this strategy on the fibrotic lung has not yet been documented. With this observational study we aim at documenting the effect of PEEP titration maneuver based on end-expiratory trans-pulmonary pressure on lung mechanics of patients with pulmonary fibrosis and UIP pattern,

ELIGIBILITY:
Inclusion Criteria:

* pulmonary fibrosis with UIP pattern
* subjected to endotracheal intubation and controlled mechanical ventilation for acute respiratory failure
* candidate to a trial of PEEP titration according to positive end expiratory pressure.

Exclusion Criteria:

* chest wall deformities
* chronic obstructive pulmonary disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung fibrosis and UIP pattern undergoing esophageal manometry and controlled mechanical ventilation for acute respiratory failure admitted to the Intensive Care Unit and Respiratory Intensive Care Unit of the University Hospital of Modena that will fulfill the eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung elastance | 2 hours.
  The effect of PEEP titration according to end-expiratory transpulmonary pressure on lung elastance will be analyzed.

SECONDARY OUTCOMES:
P/F ratio | 2 hours
  The effect of PEEP titration according to end-expiratory transpulmonary pressure on P/F ratio will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided